CLINICAL TRIAL: NCT04059523
Title: A Phase 1b, Multicenter, Open-Label, Parallel-Group, Maximal Use Systemic Exposure (MUSE) Study to Evaluate the Pharmacokinetics, Safety and Tolerability of S6G5T-3 Compared to Retin-A® 0.1% in Subjects With Moderate to Severe Acne Vulgaris
Brief Title: MUSE Study to Evaluate the Pharmacokinetics, Safety and Tolerability of S6G5T-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGT-65-03
Record Dates: First submitted 2019-08-01; First posted 2019-08-16 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S6G5T-3 (Experimental): topical cream
  Interventions: Drug: S6G5T-3
- Retin-A® 0.1% Cream (Active Comparator): topical cream
  Interventions: Drug: Retin-A® 0.1% Cream

INTERVENTIONS:
Drug: S6G5T-3 — once daily
  Arms: S6G5T-3
Drug: Retin-A® 0.1% Cream — once daily
  Arms: Retin-A® 0.1% Cream

SUMMARY:
To assess the degree of systemic exposure of S6G5T-3 compared to the Reference Listed Drug (RLD) Retin-A® 0.1% Cream when applied topically once daily for 14 days, under maximal use conditions in adolescents ≥12 years of age and adults with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 9 years of age or older.
2. Subject must consent to participate, verified by signing an approved written Informed Consent Form (ICF).
3. Subjects must be generally healthy and free from any clinically significant disease, other than acne vulgaris, that might interfere with the study evaluations
4. All females of child-bearing potential and premenarchal, excluding women who are surgically sterile

Exclusion Criteria:

1. Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne etc.) or severe acne requiring systemic treatment.
2. Underlying disease which requires the use of topical or systemic therapy which may confound study results or make results difficult to interpret.;
3. Subjects unable to communicate well with the site study team (i.e., language problem, poor mental development or impaired cerebral function).
4. Any other factor that, in the opinion of the Investigator, would prevent the subject from complying with the requirements of the protocol.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of S6G5T-3 as measured by the maximum observed plasma concentration | 14 days
  The degree of systemic exposure of S6G5T-3 compared to the Reference Listed Drug (RLD) when applied topically once daily for 14 days, under maximal use conditions in subjects with acne vulgaris. Cmax = Maximum plasma concentration will be calculated

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - DermResearch, Inc., Austin, Texas
  - J&S Studies, Inc, College Station, Texas